CLINICAL TRIAL: NCT06368414
Title: A Study of Treatment-free Remission in Chronic Phase Chronic Myeloid Leukemia in Combination With Asciminib and Tyrosine Kinase Inhibitors
Brief Title: A Study of Treatment-free Remission in Chronic Phase Chronic Myeloid Leukemia
Acronym: AsterA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Korean Society of Hematology (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCMLWP-2021-04
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Chronic Myeloid Leukemia, Chronic Phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — asciminib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Asciminib arm (Other)
  Interventions: Drug: Asciminib

INTERVENTIONS:
Drug: Asciminib — that patients who lost MR3.0 after stopping TKIs, thus failed to maintain treatment-free remission can achieve second sustainable MR4.5 by sustainable MR4.5 for more than 3 years once regained and prolong MRFS by adding asciminib to TKIs. Patients will be restarted on TKIs when they fail sustaining MR3.0 after cessation because restarting TKIs when loss of MR3.0 is reasonable in this situation

SUMMARY:
To evaluate the efficacy of asciminib adding on tyrosine-kinase inhibitors (TKI) to achieve treatment-free remission (TFR) in chronic myeloid leukemia (CML) patients in chronic phase who failed prior cessation study of TKI

DETAILED DESCRIPTION:
We expect that patients who lost MR3.0 after stopping TKIs, thus failed to maintain treatment-free remission can achieve second sustainable MR4.5 by sustainable MR4.5 for more than 3 years once regained and prolong MRFS by adding asciminib to TKIs. Patients will be restarted on TKIs when they fail sustaining MR3.0 after cessation because restarting TKIs when loss of MR3.0 is reasonable in this situation.

ELIGIBILITY:
Inclusion Criteria:

1. 19 year or older
2. CP-CML patients who are taking current TKIs (imatinib, nilotinib or dasatinib) for 5 years or more
3. Patients who have failed maintaining MR3.0 after 1 or more cessation trial of TKIs.
4. Patients who regained MR3.0 or deeper molecular response by TKIs retrial after TKI cessation failure at the time of screening
5. Taking TKIs over 12 weeks for the retrial of TKIs after TKI cessation failure
6. Patients who agree with stopping asciminib and TKIs after maintaining 23 year-duration of MR4.5
7. Adequate end organ function as defined by:

   * Total bilirubin (TBL) < 3 x upper limit of normal (ULN); patients with Gilbert's syndrome may only be included if TBL ≤ 3.0 x ULN or direct bilirubin ≤ 1.5 x ULN
   * Creatinine clearance (ClCr) ≥ 30 mL/min as calculated using Cockcroft-Gault formula
   * Serum lipase ≤ 1.5 x ULN. For serum lipase > ULN - ≤ 1.5 x ULN, value must be considered not clinically significant and not associated with risk factors for acute pancreatitis
8. Patients who can sign the informed consent of their own free will

Exclusion Criteria:

1. Patients who experienced grade 3 or higher adverse events with TKIs (imatinib, dasatinib, and nilotinib).
2. Patients who are receiving any other investigational agents.
3. Patients who currently have uncontrolled infections
4. Patients who previously received Chimeric antigen receptor T-cell (CAR-T cell) therapy, allogeneic hematopoietic stem cell transplantation (allo-HSCT) or biologic therapy.
5. Patients with clinically significant cardiovascular disease or gastrointestinal dysfunction.
6. Patients who have a history of thromboembolic episodes within 3 months prior to the study enrollment.
7. Patients with active hepatitis B or C with uncontrolled disease activity.
8. Patients who have active malignancies requiring treatment other than CML.
9. Patients with any severe and/or uncontrolled medical conditions or other conditions that could adversely impact on patients' ability to participate in the study.
10. Patients with psychiatric illness/social situations that would limit compliance with study requirements.
11. Pregnant women are excluded from this study Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with asciminib and TKIs, breastfeeding should be discontinued if the mother is treated with asciminib and TKIs.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
MR3.0 or less by 1 year | by 1 year
  To evaluate the cumulative incidence of sustained MR3.0 or less by 1 year of cessation of TKI and asciminib

CONTACTS AND LOCATIONS:
Overall Officials: Hawk Kim, Study Chair — Korean Society of Hematology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levey AS, Coresh J, Greene T, Stevens LA, Zhang YL, Hendriksen S, Kusek JW, Van Lente F; Chronic Kidney Disease Epidemiology Collaboration. Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. Ann Intern Med. 2006 Aug 15;145(4):247-54. doi: 10.7326/0003-4819-145-4-200608150-00004. PMID 16908915

DOCUMENTS (2):
  • Study Protocol (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/14/NCT06368414/Prot_000.pdf
  • Study Protocol (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/14/NCT06368414/Prot_001.pdf